CLINICAL TRIAL: NCT05087576
Title: Chinese American Family Caregiver Writing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-1547
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-09

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Helping writing (Experimental): During the first writing session, participants will be informed that people benefit from learning about other cancer caregivers' experiences, and that the first three sessions will consist of writing exercises designed to help them think about their cancer caregiving experiences and to prepare them for writing a helpful letter to other Chinese cancer caregivers during the fourth and final writing session.
  Interventions: Behavioral: Expressive Helping
- Caregiving Facts writing (Active Comparator): During each week, participants in the control group will be asked to write facts about their experience with cancer caregiving (e.g., type of treatment their loved one is receiving) and will be asked to avoid writing about their emotions. Participants in this group will be told that their writing will not be shared with others outside of the research team.
  Interventions: Behavioral: Caregiving Fact writing

INTERVENTIONS:
Behavioral: Expressive Helping — Expressive helping integrates two distinct areas of research showing that emotional disclosure over writing and support giving improves psychological well-being among healthy and clinical populations. Participants write 4 brief structured writing sessions.
  Arms: Expressive Helping writing
Behavioral: Caregiving Fact writing — Factual Writing has been used with in other writing-based interventions (e.g., expressive writing). It is also completed in 4 brief structured writing sessions.
  Arms: Caregiving Facts writing

SUMMARY:
The Chinese American Family Caregiver Writing Study is a Randomized Controlled Trial (RCT) testing the efficacy of the Expressive Helping (EH) intervention among Chinese Americans who are providing care for family members undergoing cancer treatment.

DETAILED DESCRIPTION:
Because the psychosocial health of Chinese cancer patients and their caregivers are linked, there is a need to improve health outcomes for not just the patients, but also for the caregivers. While many caregiving interventions have focused on the caregiver-patient dyad as the "the unit of care", interventions that solely target caregivers are crucial given the emotional, social, financial, and physical toll of caregiving. To address this need, investigators are testing a writing intervention, Expressive Helping (EH), with Chinese family members who are providing care for their family members diagnosed with cancer. Over four brief structured writing sessions, participants write about their cancer caregiving experiences, disclosing their emotions and providing encouragement and guidance, with the knowledge that their narratives will be shared with and used as a resource for other Chinese cancer caregivers. Participants will be adult cancer caregivers of Chinese descent. After screening and consent, eligible participants will be enrolled in a 1:1 randomized controlled trial. Assessments of psychological symptoms will occur at baseline (prior to randomization), 1-month post-intervention, and 3-month post-intervention. Investigators will also assess potential mediators and moderators of the potential intervention effects. Investigators interacting with the participants will be blind to condition assignment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Of Chinese descent
* Informal (i.e., uncompensated) caregiver of individual diagnosed with cancer

Exclusion Criteria:

* Inability to read or write English or Traditional/Simplified Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms assessed by the Center for Epidemiologic Studies Depression Scale | Baseline to 1-month follow-up and 3-month follow-up
  Depressive symptoms will be measured with the 20-item Center for Epidemiologic Studies Depression Scale (CES-D). Score ranges from 0-60, with higher scores indicating a worse outcome.
Changes in life satisfaction assessed by the Satisfaction with Life Scale. | Baseline to 1-month follow-up and 3-month follow-up
  Life satisfaction will be measured by the 5-item Satisfaction with Life Scale (SWLS). Score ranges from 5-35, with higher scores indicating a better outcome.
Changes in caregiver quality of life assessed by the Caregiver quality of life index - Cancer | Baseline to 1-month follow-up and 3-month follow-up
  Caregiver quality of life will be measured by the 35 item Caregiver quality of life index - Cancer (CQOL-C). Score ranges from 0-140, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Changes in post-traumatic growth assessed by the Post-traumatic Growth Inventory | Baseline to 1-month follow-up and 3-month follow-up
  Post-traumatic growth will be measured by the 21-item Post-traumatic Growth Inventory (PTGI). Score ranges from 0-105, with higher scores indicating a better outcome.
Changes in sleep quality assessed by the Pittsburgh Sleep Quality Index | Baseline to 1-month follow-up and 3-month follow-up
  Sleep quality will be measured by the 19-item Pittsburgh Sleep Quality Index (PSQI). Score ranges from 0-21, with higher scores indicating a worse outcome.
Changes in caregiver strain assessed by the Zarit Burden Interview | Baseline to 1-month follow-up and 3-month follow-up
  Caregiver strain will be measured by the 22-item Zarit Burden Interview. Score ranges from 0-88, with higher scores indicating a worse outcome.
Changes in intrusive thoughts assessed by the Impact of Event scale. | Baseline to 1-month follow-up and 3-month follow-up
  Intrusive thoughts will be measured by the 15 item Impact of Event scale (IES). Score ranges from 0-40, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All IPD will be protected and maintained by the study team